CLINICAL TRIAL: NCT07313098
Title: Longitudinal Assessment of Protein Markers in the Cerebrospinal Fluid of Patients With Central Nervous System Involvement
Acronym: HJ-COLOCS
Status: Not yet recruiting | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HJ-23-HJ-COLOCS
Record Dates: First submitted 2025-11-18; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Neurologic Disorder; Central Nervous System Diseases
Keywords: Cerebrospinal Fluid; Central Nervous System Diseases; Neurologic Disorder
MeSH Terms: conditions — Nervous System Diseases; Central Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Leftover cerebrospinal fluid from medical procedures, residual blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Patients with a neurological condition diagnosed by a physician and requiring CSF sampling as part of their routine care

SUMMARY:
In the context of adult pathology, research into biomarkers in cerebrospinal fluid (CSF) has already identified proteins that are commonly used for the early diagnosis of certain neurodegenerative diseases. However, the lack of data available in the literature on pediatric diseases has limited the use of biomarkers in routine practice in children. Importantly, our group has pioneered the establishment of CSF biomarkers in children (e.g., measurement of interferon alpha in CSF by ultra-sensitive digital ELISA), which will undoubtedly be used in routine clinical practice in the future. In light of these arguments, the establishment of a CSF biobank will have major clinical implications, given the rarity of the diseases treated and the number of patients followed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a neurological condition diagnosed by a physician requiring cerebrospinal fluid (CSF) collection, through:

   * Neurosurgical procedure (EVD, VP shunt, VSG shunt, tumor surgery, spinal surgery with dural opening, ELD);
   * Lumbar puncture (LP).
2. Patients who have (or whose legal guardians, where applicable, have) consented to the storage and reuse of residual biological samples collected during the course of care within the biological collection.

Exclusion Criteria:

1. Objection by the patient and/or the legal guardian, if the patient is a minor, to participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a neurological condition diagnosed by a physician requiring cerebrospinal fluid (CSF) collection as a part of their health care
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2036-01-01 (Estimated); Study Completion 2036-01-01 (Estimated)

PRIMARY OUTCOMES:
Longitudinal evolution of protein markers in CSF from patients with central nervous system involvement | 2021 - 2035

SECONDARY OUTCOMES:
Longitudinal changes in inflammatory protein levels in the CSF of patients with post-hemorrhagic hydrocephalus | 2021 - 2035
Proteomic characterization of several neuroinflammatory diseases | 2021 - 2035
Identification of biomarkers of severity in children with traumatic brain injury | 2021 - 2035
Comparison of CSF biomarkers with data generated in serum (when available) | 2021 - 2035
  Proteomic analysis by comparing LCS biomarker results with data generated in serum, in order to discover new biomarkers relevant to the pathology under study.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Louise FREMOND, Pr, MD, Principal Investigator — Imagine Institute
Locations (1):
- Hôpital Necker-Enfants malades, Paris, France